CLINICAL TRIAL: NCT05333016
Title: A Dyadic Approach to Cancer Care: a Feasibility and Efficacy Partner-based Exercise Study
Acronym: C4C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Melanie Keats, Affiliated Scientist, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NSH Caring 4 Cancer Caregivers
Record Dates: First submitted 2022-04-04; First posted 2022-04-18 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Cancer
Keywords: Cancer; Caregiver burden; Survivor; Dyad; Exercise; Intervention; Feasibility
MeSH Terms: conditions — Neoplasms; Caregiver Burden; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multimodal Exercise Intervention (Experimental): 12-week, twice weekly partner-based multimodal exercise program
  Interventions: Behavioral: Multimodal exercise

INTERVENTIONS:
Behavioral: Multimodal exercise — Multimodal exercise programming including aerobic, resistance, balance, and flexibility exercises

SUMMARY:
The primary goal of this study will be to assess the feasibility and acceptability of a partner-based 12-week exercise intervention for cancer caregivers and their care recipient. The researchers will also explore the preliminary effectiveness of the exercise program on caregiver burden and physical and psychological health of both the family caregiver and the care recipient.

DETAILED DESCRIPTION:
NEED: Cancer has been characterized as a family affair, as it is a disease in which both the patient and their family members are confronted by considerable physical and psychological stressors. With an anticipated 80% increase in the average number of new cancer diagnoses by 2030 and rapidly escalating health care costs, there has been a shift to outpatient and home-based care. In doing so, family members are increasingly being called upon to participate as informal caregivers (i.e., an individual who provided uncompensated care). Despite being a key partner in the supportive care of the cancer patient, family caregivers are often inadequately prepared or supported to take on this critical role, subsequently putting their own health and well-being at risk and by extension, that of the cancer patient/survivor. Preliminary data suggests that exercise interventions show promise in mitigating caregiver burden and improving health outcomes for both the caregiver and the patient/survivor. To date, however only two studies have examined the benefit of exercise interventions on family caregiver and patient outcomes within the cancer care context.

GOAL: The primary goal of this study will be to assess the feasibility and acceptability of a partner-based 12-week exercise intervention. The investigators will also explore the preliminary effectiveness of the exercise program on caregiver burden and physical and psychological health of both the family caregiver and the care recipient.

WHO: Participants will include adult primary caregivers and cancer patients/survivors of all cancers and stages at any point along the cancer care trajectory.

HOW: Using both surveys and participant interviews, the participant experience and impact (e.g., physical and psychological health benefits) of a 12-week, partner-based exercise intervention will be evaluated. The 12-week exercise program will include a combination of aerobic, resistance, balance, and flexibility exercises delivered in a partner-based setting twice weekly at a dedicated cancer and exercise lab.

ELIGIBILITY:
Inclusion Criteria (all):

* 18+ years
* able to perform discontinuous low intensity physical activity at a minimum
* able to provide informed written consent in English.

Inclusion Criteria (cancer patients/survivors)

- are along any stage of the cancer continuum (i.e., pre-treatment, receiving active treatment, and up to 5 years post-treatment)

Inclusion Criteria (informal caregivers)

* must be currently providing physical and/or psychological support to an adult (+18 years) cancer patient/survivor
* not be exceeding current Canadian physical activity guidelines (i.e., 150 minutes of moderate-to-vigorous physical activity per week)

Exclusion Criteria (all):

- Patients/survivors and caregivers will be excluded from the study if they have any medical conditions that would contraindicate exercise

Exclusion Criteria (informal caregivers)

- Bereaved caregivers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Recruitment | Through study completion, about 2 years
  Participant accrual as defined as the number of eligible participant dyads who consents to participate
Intervention Adherence | Through study completion, about 2 years
  Participant program adherence calculated as percentage of exercise sessions completed divided by total number of available exercise sessions over 12-week intervention
Adverse Events | Through study completion, about 2 years
  Adverse and serious adverse events will be recorded
Attrition | Through study completion, about 2 years
  Participant attrition calculated as percentage of patients who complete 12-week study divided by number who withdraw from study
Participant Satisfaction | Post intervention, about 12-weeks after baseline
  Participant satisfaction will be assessed by semi-structured interviews (no min/max)

SECONDARY OUTCOMES:
Caregiver Burden | Pre to post intervention (12-week change)
  Assessed by the 22-item Zarit Burden Interview (ZBI). Responses are scored on a 5-point Likert scale ranging from 0 (never) to 4 (nearly always) with the sum of scores ranging from 0 to 88 (higher scores indicate higher burden)
Body Mass Index (BMI) | Pre to post intervention (12-week change)
  Weight (kg) and height (m) will be used to calculate BMI
Body Composition | Pre to post intervention (12-week change)
  Waist and hip circumference
Resting heart rate | Pre to post intervention (12-week change)
  Resting heart rate
Resting Blood Pressure | Pre to post intervention (12-week change)
  Resting systolic and diastolic blood pressure
Aerobic Fitness | Pre to post intervention (12-week change)
  The 6-minute walk test will be used to assess aerobic capacity
Upper Body Strength | Pre to post intervention (12-week change)
  Grip strength will be measured using a hand-held dynamometer
Muscular Endurance | Pre to post intervention (12-week change)
  Lower body muscular endurance will be assessed using the 30-second sit-to-stand
Balance | Pre to post intervention (12-week change)
  Balance will be assessed using the one-legged stance
Flexibility | Pre to post intervention (12-week change)
  Flexibility will be assessed using the sit-and-reach and shoulder flexibility
Caregiver Quality of Life | Pre to post intervention (12-week change)
  Quality of life will be assessed using the Short-Form Health Survey- SF-36. The SF-36 consists of 36 questions that cover 8 health domains/subscales (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health). The total scale score ranges from 0 to 100 with higher values representing higher quality of life.
Cancer Patient Quality of Life | Pre to post intervention (12-week change)
  Quality of life for cancer patients will be assessed using the Functional Assessment of Cancer Therapy - General survey. The combined 27-item scale provides subscale scores physical (7-items), functional (7-items), emotional (6-items), and social/family (7-items) well-being. The sum of scores on the five domains evaluates a participants' quality of life with higher scores (ranging from 0-108) denoting higher quality of life.
Cancer Patient Fatigue | Pre to post intervention (12-week change)
  Fatigue will be assessed using the 13-item Functional Assessment of Chronic Illness Therapy - Fatigue survey. Scores range from 0-52 with higher scores indicating better functioning/less fatigue
Self-Reported Physical Activity | Pre to post intervention (12-week change)
  Physical activity will be assessed using the Godin Leisure Time Exercise Questionnaire. Total score ranges from 0 to no maximum.
General Health (EuroQol) 5 Dimension - 5 Level | Pre to post intervention (12-week change)
  Mobility, self-care, usual activities, pain/discomfort, anxiety/depression (EuroQol-5Dimension-5Level; EQ-5D-5L); higher scores indicate higher problems (range 0-1)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Keats, PhD, Principal Investigator — Dalhousie University / Nova Scotia Health
Locations (1):
- Physical Activity and Cancer (PAC) Lab, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Physical Activity and Cancer Lab website — http://www.thepaclab.com